CLINICAL TRIAL: NCT00331526
Title: Phase II Trial of Intralesional Adoptive Cellular Therapy of Glioblastoma With Interleukin-2-Stimulated Lymphocytes
Brief Title: Cellular Adoptive Immunotherapy in Treating Patients With Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000471241; HOAG-CBRG-98-09
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult gliosarcoma; adult giant cell glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — aldesleukin; Chemotherapy, Adjuvant

INTERVENTIONS:
Biological: aldesleukin
Biological: therapeutic autologous lymphocytes
Procedure: adjuvant therapy
Procedure: conventional surgery

SUMMARY:
RATIONALE: Biological therapies, such as cellular adoptive immunotherapy, may stimulate the immune system in different ways and stop tumor cells from growing. Aldesleukin may stimulate the white blood cells, including lymphokine-activated killer cells, to kill tumor cells. Giving cellular adoptive immunotherapy during or after surgery may kill more tumor cells.

PURPOSE: This phase II trial is studying how well cellular adoptive immunotherapy works in treating patients with glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility, side effects, and toxicity associated with intracranial cellular adoptive immunotherapy comprising aldesleukin-stimulated lymphokine-activated killer cells in patients with glioblastoma multiforme.
* Determine progression-free and overall survival of these patients.
* Compare survival of these patients to that of contemporary and historical controls.

OUTLINE: Patients undergo therapeutic craniotomy.

Patients undergo leukapheresis to obtain lymphokine-activated killer (LAK) cells 3-7 days before therapeutic craniotomy OR 4-6 weeks after therapeutic craniotomy. Patients receive cellular adoptive immunotherapy comprising aldesleukin-stimulated LAK cells intracranially at the time of therapeutic craniotomy OR via an Ommaya reservoir (placed during craniotomy) no sooner than 4-6 weeks after therapeutic craniotomy.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of primary malignant glioblastoma multiforme (i.e., grade IV anaplastic astrocytoma)
* Primary treatment (surgery, radiation, and/or chemotherapy) has been completed
* Candidate for surgery and willing to undergo craniotomy
* No progressive or recurrent disease
* No residual disease that requires reoperation, additional gamma therapy, or other modality

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 70-100% (i.e., if symptomatic, bedridden < half of a waking day)
* Life expectancy ≥ 2 months
* Not pregnant
* Negative pregnancy test
* U.S. residents only
* No hematopoietic, hepatic, renal, cardiovascular, or pulmonary laboratory values or other medical circumstances that would preclude surgery or aldesleukin therapy
* No serious concurrent medical or psychiatric illness that would preclude informed consent or study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior anticancer therapy and recovered
* Prior stereotactic or gamma knife radiosurgery allowed

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 1999-02; Primary Completion 2008-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Side effects and toxicity
Progression-free survival and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Robert O. Dillman, MD, FACP, Study Chair — Hoag Memorial Hospital Presbyterian
Locations (1):
- Hoag Cancer Center at Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States

REFERENCES:
- [Result] Dillman RO, Duma CM, Ellis RA, Cornforth AN, Schiltz PM, Sharp SL, DePriest MC. Intralesional lymphokine-activated killer cells as adjuvant therapy for primary glioblastoma. J Immunother. 2009 Nov-Dec;32(9):914-9. doi: 10.1097/CJI.0b013e3181b2910f. PMID 19816190